CLINICAL TRIAL: NCT02999204
Title: Effect of Vitamin D3 Supplementation on Arterial and Bone Remodeling in Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Mark L. Lipman, Associate Professor of Medicine, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #10-010
Record Dates: First submitted 2016-08-29; First posted 2016-12-21 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Renal Insufficiency, Chronic; Vascular Stiffness; Bone Diseases, Metabolic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 5,000 units per week (Active Comparator): Patient receive a dose that is considered within the standard dosing range for Vitamin D3 for one year.
  Interventions: Drug: Vitamin D3
- Vitamin D3 50,000 units per week (Experimental): Patients receive a more aggressive Vitamin D3 dosing regimen of 50,000 units weekly for the first 3 months. At this point Vitamin D3 levels are measured. If the patient is Vitamin D3 replete (>75 nmol/L) then the dose is reduced to the equivalent of 25,000 units per week for the next 9 months. If the level is below this threshold then 50,000 units per week is continued for the next 9 months
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Two different doses of Vitamin D3
  Other Names: cholecalciferol

SUMMARY:
To evaluate in patients with chronic kidney disease the impact of two dosages of per os vitamin D3 supplementation (cholecalciferol) on large arterial stiffness (evaluated non invasively by pulse wave velocity and high-resolution echotracking system). We will also study arterial calcification (lateral abdominal radiography and echocardiogram), arterial remodeling (high-resolution echotracking system), endothelial function (evaluated by a non-invasive finger biosensor device), and bone remodeling (evaluated by serum biomarkers and bone mineral density).

DETAILED DESCRIPTION:
Structural changes to large arteries and abnormalities in mineral and bone metabolism are frequent manifestations in patients with chronic kidney disease (CKD). Together, they contribute in a large part to the heightened morbidity and mortality observed in this population.

Epidemiological data in end stage renal disease and in the general population suggest the existence of a bone-vascular axis. Metabolic bone disease (MBD) in CKD encompasses altered bone remodeling and the propensity for vascular calcification. These pathological processes are driven by the multiple disorders of mineral metabolism in CKD, among them, abnormalities of vitamin D metabolism.

Vitamin D deficiency [25(OH)D] is widely observed in CKD patients and has been associated with an increased rate of cardiovascular events in both the general population and in CKD patients. The mechanisms involved are not clearly established. Vitamin D influences blood pressure through effects on the renin-angiotensin system (via a vitamin D response element in the renin gene), vascular smooth muscle cells and cardiomyocyte proliferation and hypertrophy, vascular inflammation and calcification. Vitamin D deficiency has been associated with large arterial stiffness in end-stage renal disease patients. Aortic and carotid stiffness are independent predictors of cardiovascular and overall mortality in end-stage renal disease patients. Large arterial remodeling and stiffening could be the missing pathogenic link between vitamin D deficiency and increased cardiovascular event rate.

In terms of mineral metabolism, many CKD patients develop secondary hyperparathyroidism. This results from a combination of hyperphosphatemia, hypocalcemia and low levels of active Vitamin D [1,25(OH)D2]. Since several observational studies have shown that parathyroid hormone (PTH) levels are inversely correlated with blood 25(OH)D levels, it is possible that 25(OH)D deficiency may also be contributing to the hyperparathyroid state. Secondary hyperparathyroidism contributes to cardiovascular risk and to bone disease. Elevated PTH has been associated with large arterial stiffness and remodeling. Elevated PTH is also associated with high bone turnover and participates in the development of bone disease of CKD-MBD. Bone disease in CKD-MBD comprises abnormalities in bone turnover, mineralization, linear growth and strength. Bone biopsy remains the gold standard for evaluation of bone disease in CKD but its invasive nature limits its practice. Serum biomarkers of bone remodeling allow direct estimation of bone remodeling but lack evaluation and precision. Among them, guidelines issued by Kidney Disease Improving Global Outcomes (KDIGO) recommend PTH (1-84) and bone specific alkaline phosphatase (BSALP). Other biomarkers exist including osteocalcin, osteoprotegerin, tartrate-resistant acid phosphate-5b (TRAP-5b), pyridinoline and deoxypyridinoline, procollagen type 1 amino-terminal extension peptides, C terminal cross-link (CTX) , FGF-23 and fetuin-A. The major limitation of the use of these biomarkers is their kidney-dependent elimination that affects their measured levels depending on the degree of kidney dysfunction. We have chosen to study, in addition to PTH (1-84) and BSALP, CTX, osteoprotegerin, osteocalcin, fetuin-A and fibroblast growth factor-23 (FGF-23) because a relationship between these biomarkers and arterial disease has never been demonstrated.

This study seeks to compare the impact of standard versus aggressive Vitamin D3 supplementation (in Vitamin D deficient CKD patients) on important vascular and bone health endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage 3-4 [estimated glomerular filtration rate (GFR) by modification of diet in renal disease (MDRD) formula between 15 and 60 ml/min/1.73m2].
* Serum vitamin D level<50 nmol/L.

Exclusion Criteria:

* Patient with estimated GFR by MDRD formula below 15 or above 60 ml/min/1.73m2).
* Serum vitamin D level >50 nmol/L.
* Liver disease manifested by elevated alanine aminotransferase (ALT) more than 3 times the upper limit of normal reference range, elevated gamma-glutamyl transferase (GGT) and total bilirubin levels.
* History of malabsorption or chronic diarrhea.
* Patients on biphosphonates, estrogen replacement therapy, PTH analogs, glucocorticosteroids, calcimimetics, and active vitamin D [1,25(OH)].
* Patients on antiepileptic medications or other medications affecting vitamin D metabolism (e.g. phenobarbital, phenytoin, rifampicin).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Aortic stiffness evaluated by pulse wave velocity (PWV) (Sphygmocor ® ) | 12 months
  Parameter measured in meters per second.

SECONDARY OUTCOMES:
Carotid stiffness evaluated by high resolution echotracking system (Art-lab®). | 12 months
  Parameter measured as the difference in millimeters in carotid artery diameter between systole and diastole.
Endothelial function evaluated by Endo-PAT2000® system | 12 months
  Parameter measured as the reactive hyperemia index as calculated by the Endo-PAT2000® system software.
Aortic valve calcification obtained from echocardiography. | 12 months
  Parameter measured using a semi-quantitative scoring system based on scale of 1-4 as described by Rosenhek et al, New England Journal of Medicine 2000;343 (9):611.
  1-no calcification, 2-mildly calcified (small isolated spots), 3-moderately calcified (multiple larger spots), 4-heavily calcified (extensive thickening and calcification of all cusps).
Calcification of the aorta obtained by plain lateral radiography. | 12 months
  Parameter measured using a semi-quantitative scoring system based on a scale of 0-3 as described by Kauppila et al, Atherosclerosis 1997;132:245.
  0-no calcification, 1-small scattered calcific deposits filling less than 1/3 of the longitudinal wall of the aorta, 2-one third or more, but less than two thirds of the longitudinal wall of the aorta calcified, 3-two thirds or more of the longitudinal wall of the aorta calcified.
Bone mineral density | 12 months
  Osteodensitometry of the lumbar spine, hip, and distal radius, using dual-energy X-ray absorptiometry and reported in grams per square centimeter.
Parathyroid hormone levels | 12 months
  Measurement of parathyroid hormone levels using a commercially available intact parathyroid hormone ELISA kit with values reported in ng/L.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Lipman, M.D., Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guerin AP, Blacher J, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness attenuation on survival of patients in end-stage renal failure. Circulation. 2001 Feb 20;103(7):987-92. doi: 10.1161/01.cir.103.7.987. PMID 11181474
- [Result] London GM, Guerin AP, Verbeke FH, Pannier B, Boutouyrie P, Marchais SJ, Metivier F. Mineral metabolism and arterial functions in end-stage renal disease: potential role of 25-hydroxyvitamin D deficiency. J Am Soc Nephrol. 2007 Feb;18(2):613-20. doi: 10.1681/ASN.2006060573. Epub 2007 Jan 3. PMID 17202417
- [Result] Kendrick J, Targher G, Smits G, Chonchol M. 25-Hydroxyvitamin D deficiency is independently associated with cardiovascular disease in the Third National Health and Nutrition Examination Survey. Atherosclerosis. 2009 Jul;205(1):255-60. doi: 10.1016/j.atherosclerosis.2008.10.033. Epub 2008 Nov 11. PMID 19091317
- [Result] Motiwala SR, Wang TJ. Vitamin D and cardiovascular disease. Curr Opin Nephrol Hypertens. 2011 Jul;20(4):345-53. doi: 10.1097/MNH.0b013e3283474985. PMID 21519252
- [Result] Artaza JN, Mehrotra R, Norris KC. Vitamin D and the cardiovascular system. Clin J Am Soc Nephrol. 2009 Sep;4(9):1515-22. doi: 10.2215/CJN.02260409. Epub 2009 Aug 20. PMID 19696220
- [Result] Barreto DV, Barreto FC, Liabeuf S, Temmar M, Boitte F, Choukroun G, Fournier A, Massy ZA. Vitamin D affects survival independently of vascular calcification in chronic kidney disease. Clin J Am Soc Nephrol. 2009 Jun;4(6):1128-35. doi: 10.2215/CJN.00260109. Epub 2009 May 14. PMID 19443628